CLINICAL TRIAL: NCT03036683
Title: The Effect of Transcranial Direct Current Stimulation on Risk-taking and Aggression in Offenders
Brief Title: Transcranial Direct Current Stimulation in Offenders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Olivia Choy (Other)
Collaborators: RWTH Aachen University (Other)
Responsible Party: Sponsor-Investigator, Olivia Choy, PhD candidate, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: EK 341/16
Record Dates: First submitted 2017-01-26; First posted 2017-01-30 (Estimated); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Aggression; Risk-Taking; Antisocial Behavior
MeSH Terms: conditions — Aggression; Risk-Taking; Antisocial Personality Disorder | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anodal stimulation (Experimental): Participants in the active stimulation group will undergo anodal transcranial direct current stimulation (tDCS). tDCS will be delivered by a battery-driven, constant-current stimulator connected to two saline-soaked surface sponge electrodes. An anodal electrode (25cm2) will be placed over the right dorsolateral prefrontal cortex and one cathodal electrode (100cm2) will be placed over the left supraorbital area at least 5cm from the anode. Scalp electrodes will be positioned according to the 10-20 EEG international system. A current of 2mA will be applied for 20 minutes and the current will be ramped up and down over 20 seconds at the beginning and end of the stimulation period.
  Interventions: Device: Transcranial direct current stimulation
- Sham stimulation (Sham Comparator): The sham tDCS condition will involve the same placement of the electrodes, current intensity, and ramp-up/down time as the active tDCS condition, but stimulation will only last for 30 seconds.
  Interventions: Device: Sham transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — Transcranial direct current stimulation will be administered for 20 minutes using a CE approved stimulator (NeuroConn, Ilmenau, Germany).
  Arms: Anodal stimulation
Device: Sham transcranial direct current stimulation — The same device will be used as in the active stimulation group, but stimulation will be terminated after 30 seconds.
  Arms: Sham stimulation

SUMMARY:
This study investigates the effect of upregulating prefrontal cortex activity on risk-taking, and antisocial and aggressive behavior in violent offenders. In the double-blind, randomized controlled trial, using a within-subject crossover design, each participant will undergo anodal transcranial direct current stimulation of the right dorsolateral prefrontal cortex and sham stimulation. After each stimulation session, neural activity and behavioral responses to tasks assessing risk-taking and aggressive behavior will be recorded. The effect of tDCS on violent offenders will also be assessed in comparison to age and gender-matched healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 50 years of age
* Able to understand the nature of the study and give informed consent
* Individuals in the violent offender group must have a record of repeated violent criminal offending (at least 2 felonies).
* Individuals in the violent offender group must have been convicted solely due to crimes involving violence motivated by impulsive aggression.

Exclusion Criteria:

* Presence of any contraindications for functional magnetic resonance imaging (fMRI)
* History of significant medical illness
* History of any neurological condition
* Diagnosis of schizophrenia
* History of epilepsy
* Head injury
* Mental retardation

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Number of balloon pumps in the Balloon Analogue Risk Task after stimulation | Within 1 hour after the 20-minute tDCS or sham session ends
  The number of balloon pumps, measured by the number of times subjects press a button to pump up a computerized balloon over 60 trials, will be assessed.
Neural activity during Balloon Analogue Risk Task after stimulation | Within 1 hour after the 20-minute tDCS or sham session ends
  Functional brain activity and connectivity will be assessed using functional magnetic resonance imaging.
Aggressive behavior after stimulation | Within 1 hour after the 20-minute tDCS or sham session ends
  This will be assessed according to performance on the violent video game, Carmageddon: TDR 2000 (Klasen et al., 2013; Torus Games, Bayswater, Australia, 2000) in comparison to a modified non-violent version of the game.
Neural activity during aggression task after stimulation | Within 1 hour after the 20-minute tDCS or sham session ends
  Functional brain activity and connectivity during participation in the video game will be assessed using functional magnetic resonance imaging.
Antisocial behavior inclinations after stimulation | Within 1 hour after the 20-minute tDCS or sham session ends
  This will be assessed using 8 hypothetical scenarios in which someone commits a criminal or antisocial act. Participants will respond to the likelihood that they would commit the act in the scenario according to a 10-point Likert scale.

SECONDARY OUTCOMES:
Number of participants with adverse events | Within 1 hour after the 20-minute tDCS or sham session ends
  The number of participants reporting the experience of sensations resulting from tDCS will be recorded.
Ratings of guilt or shame regarding antisocial acts after stimulation | Within 1 hour after the 20-minute tDCS or sham session ends
  This will be assessed using 8 hypothetical scenarios in which someone commits a criminal or antisocial act. Participants will respond to the likelihood that they would feel a sense of guilt or shame according to a 10-point Likert scale.
Ratings of moral wrongfulness regarding antisocial acts after stimulation | Within 1 hour after the 20-minute tDCS or sham session ends
  This will be assessed using 8 hypothetical scenarios in which someone commits a criminal or antisocial act. Participants will rate the moral wrongfulness of the acts according to a 10-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Ute Habel, PhD, Principal Investigator — RWTH Aachen University
Locations (1):
- Uniklinik RWTH Aachen, Aachen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klasen M, Zvyagintsev M, Schwenzer M, Mathiak KA, Sarkheil P, Weber R, Mathiak K. Quetiapine modulates functional connectivity in brain aggression networks. Neuroimage. 2013 Jul 15;75:20-26. doi: 10.1016/j.neuroimage.2013.02.053. Epub 2013 Mar 7. PMID 23501053